CLINICAL TRIAL: NCT06311279
Title: End to End Versus Side to End Anastomosis After Anterior Resection of Cancer Rectum
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Nabil Abdelnaser Al-ameer, assistant lecturer, physician and MD candidate, Sohag University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Soh-Med-24-03-01MD
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Rectum Cancer
Keywords: cancer rectum; Anastomosis; End to end; side to end
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Comparison between end to end and side to end anastomosis after anterior resection of cancer rectum and compare the outcomes of both surgical techniques. The main outcomes were bowel functional outcomes and QoL. Bowel functional outcomes mainly included three indexes: stool frequency, urgency, incomplete defecation, and incontinence. The secondary outcomes were surgical outcomes including operative time, postoperative hospital stay, postoperative complications, reoperation, and mortality
Who Masked: Participant, Outcomes Assessor
Masking Description: randomized comparative clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): the first group included patients who will have anterior resection with end-to-end anastomosis
  Interventions: Procedure: Anterior resection of Rectal cancer
- Group B (Active Comparator): the second group included patients will have anterior resection with side to end anastomosis.
  Interventions: Procedure: Anterior resection of Rectal cancer

INTERVENTIONS:
Procedure: Anterior resection of Rectal cancer — Anterior resection of cancer rectum and type of anastomosis (End to end or side to end)

SUMMARY:
Comparison between end to end and side to end anastomosis after anterior resection of cancer rectum and compare the outcomes of both surgical techniques. The main outcomes were bowel functional outcomes and QoL. Bowel functional outcomes mainly included three indexes: stool frequency, urgency, incomplete defecation, and incontinence. The secondary outcomes were surgical outcomes including operative time, postoperative hospital stay, postoperative complications, reoperation, and mortality.

DETAILED DESCRIPTION:
During the past two decades, remarkable progress has been made in the treatment of rectal cancer. The main goal of rectal surgery for malignancy is oncologic radicality in an effort to achieve the preservation of sphincters and sexual-urinary function.The introduction of circular stapling devices is largely responsible for their increasing popularity and utilization. Sphincter-saving procedures associated to partial or total mesorectal excision (TME) for the treatment of mid and distal rectal cancer have become increasingly prevalent as their safety and efficacy have been proved. Total mesorectal excision (TME) is the best available treatment for rectal cancer. With the advancement of surgical techniques, the majority of patients with mid and upper rectal cancer can undergo a sphincter-saving TME procedure. After TME, the most widely used reconstructive technique is straight coloanal anastomosis. With the advancement of surgical technique, the local recurrence rate after rectal cancer surgery has been decreased from 25-50% to 3-8%. Naturally, it is time to focus on how to improve bowel functional outcomes and quality of life (QoL) for rectal cancer patients. However, because the sigmoid colon is usually excised during surgery which decreases the storage volume of stool, there is a common problem seriously influencing the life quality of patients, including increased tool frequency, urgency and incontinence, which is termed as anterior resection syndrome (ARS). About 19-56% of patients would suffer from ARS. Thus, the demand for a technique with better functional outcomes made surgeons modify the straight anastomotic technique. Thus, another modified anastomotic technique, side-to-end anastomosis, which has been used since 1966, has gained attention. Side-to-end anastomosis usually needs a 3-5 cm-long colonic segment. Multiple studies on the literature have shown that compared with straight anastomosis, side-to-end anastomosis has advantages in bowel functional and operative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age to 80 years.
* Laparoscopic or open anterior resection of cancer rectum.

Exclusion Criteria:

* synchronous colorectal carcinoma
* emergency surgery
* history of colon or rectal segmental resections
* fixed rectal carcinoma who received preoperative radiotherapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-03-20 (Estimated)

PRIMARY OUTCOMES:
Operative time | Immediate postoperative
  in minutes
Anastomotic leakage | 2 weeks postoperative
  yes or No
hospital stay | 2 weeks postoperative
  in days
Mortality | 4 weeks postoperative
  yes or no
Anastomotic leak amount | 2 weeks postoperative
  in cubic centimeters

CONTACTS AND LOCATIONS:
Overall Officials: AbdElhafez H Mohamed, MD, Study Chair — Sohag University; Ahmed A Ahmed, MD, Study Director — Ain Shams University; Nabil A Al-Ameer, MD, Principal Investigator — Sohag University; Emad G Mohamed, MD, Study Director — Sohag University
Locations (1):
- Sohag university, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No